CLINICAL TRIAL: NCT01018615
Title: Steady-State Pharmacokinetic Interactions of Green Tea Catechins and Silymarin Flavonolignans in Treatment Naïve Patients With Chronic Hepatitis C Infection
Brief Title: Safety, Metabolism, and Antioxidant Activity of Silymarin and Green Tea Extract in Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-1631; R21AT003892-01A2 (NIH); CTRC-2779 (Other: University of North Carolinat at Chapel Hill)
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2014-06

CONDITIONS: Chronic Hepatitis C; Oxidative Stress
Keywords: chronic hepatitis C; silymarin; green tea catechins; green tea extract; pharmacokinetics; antioxidant activity
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Silymarin; milk-thistle extract; Tea; epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low dose silymarin and low dose EGCG (Experimental)
  Interventions: Drug: silymarin; Dietary Supplement: green tea extract (EGCG)
- high dose silymarin and low dose EGCG (Experimental)
  Interventions: Drug: silymarin; Dietary Supplement: green tea extract (EGCG)

INTERVENTIONS:
Drug: silymarin — capsules, 700 mg, twice daily, 12 days
  Other Names: milk thistle
Dietary Supplement: green tea extract (EGCG) — capsules, 196.5 mg, twice daily, 12 days
  Other Names: green tea catechins; EGCG

SUMMARY:
The purpose of this study is to determine if the safety, metabolism, and antioxidant activity of silymarin and green tea extract are changed when they are given in combination to patients with chronic hepatitis C infection.

DETAILED DESCRIPTION:
Silymarin and green tea are the two most widely used botanical products used by patients with chronic hepatitis C virus (HCV) infection. A major limitation of prior clinical investigations that may account for lack of efficacy is their use of inadequate customary oral dose regimens. Ongoing Phase II studies utilizing higher than customary doses of silymarin are based on potential disease modifying effects resulting from the potent antioxidant properties of silymarin flavonolignans. Since patients often use more than one herbal product to self-treat their disease, the use of higher than customary doses of silymarin may change silymarin's potential for herbal-herbal interactions. Pharmacokinetic interactions between silymarin and green tea catechins may change their safety/tolerability profiles, and may increase their antioxidant effects through additive or synergistic pharmacodynamic interactions. The objective of this double blind, active placebo controlled, randomized clinical trial is to characterize the pharmacokinetics and to evaluate the safety, tolerability, and antioxidant effects of an herbal cocktail consisting of silymarin and epigallocatechin gallate (EGCG) standardized green tea extract in treatment-naïve patients with chronic HCV infection. This investigation will include two treatment arms that will enroll 15 subjects per arm. Subjects will be randomized to receive in a fixed sequence either: 1) 196.5 mg EGCG followed by the coadministration of 700 mg silymarin; or 2) 700 mg silymarin followed by the coadministration of 196.5 mg EGCG. Each dosing regimen will be administered p.o. every 12 hrs for 12 days. No treatment arm uses high doses for both silymarin and EGCG in a sequence. Depending on the treatment arm, pharmacokinetic studies will be performed on plasma concentrations for six major silymarin flavonolignans and for the green tea catechin, EGCG at the end of 12 days of either silymarin or green tea extract monotherapy (Period 1), and then again after 12 days of silymarin and green tea extract given in combination (Period 2). For each treatment arm, plasma 8F2α-isoprostane concentrations, a measure of oxidative stress, will also be determined at baseline, during each period, and then at follow-up. The results from this investigation will be used to identify doses of silymarin and green tea that can be used together safely for future efficacy trials in patients with different chronic liver diseases.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for enrollment in this study if they meet the following criteria:

* Males or females; age at least 18 years at screening
* Negative urine pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of silymarin. Females of childbearing potential must be using two reliable forms of effective contraception during the study (while on drug and during follow-up)
* Hepatitis C virus (HCV) patients
* Any HCV genotype
* Never been treated or received less than 50% of standard peg-interferon-based therapy.
* No interferon-based therapy in the previous 6 months
* Serum HCV RNA above quantifiable level of detection by the assay, within 1 year of screening.
* Before entering the study, subjects must agree not to consume alcohol for 48 hours prior to PK sampling days or while on study.

Exclusion Criteria:

Subjects with any of the following will not be eligible for participation:

* Use of other milk thistle or green tea preparations within 30 days of Study Visit 1 (Day 1)
* Use of other antioxidants such as vitamin E, vitamin C, glutathione, alpha-tocopherol, within 30 days of Study Visit 1 (Day 1). A multivitamin at standard doses will be allowed.
* Use of diets containing > 6 servings per day, or 4-6 servings per day from > 8 of the vegetables and fruits listed in Appendix 2.
* Allergy/sensitivity to milk thistle, green tea or their preparations
* Inability to tolerate milk products (lactose intolerant)
* Use of any interferon-based therapy in the last 6 months.
* Use of warfarin, metronidazole or chronic use of acetaminophen greater than two grams per day
* Previous liver biopsy that demonstrated presence of cirrhosis or previous liver biopsy that demonstrated greater than or equal to 15% steatosis or evidence of steatohepatitis
* Positive test for anti-HIV or HBsAg within 3 years of screening
* Positive urine drug screen for drugs of abuse at screening
* Alcohol consumption of more than one drink or equivalent (>12 grams) per day. Patients who consumed more than this in the past must have maintained a level 12 grams or less per day of alcohol consumption for at least six months prior to screening.
* History of other chronic liver disease, including metabolic diseases, documented by appropriate test(s)
* Women with ongoing pregnancy or breast-feeding, or contemplating pregnancy
* Platelet count <130,000 cells/mm3.
* Creatinine clearance ≤30cc/min or currently on dialysis. Creatinine clearance will be calculated according to Cockcroft-Gault.
* Evidence of alcohol or drug abuse within 6 months prior to screening
* Evidence of decompensated liver disease defined as any of the following: serum albumin <3.2 g/dl, total bilirubin > 1.5 mg/dl, or PT/INR > 1.3 times normal at screening, or history or presence of ascites or encephalopathy, or bleeding from esophageal varices
* History of inflammatory bowel disease or autoimmune hepatitis
* History of solid organ or bone marrow transplantation
* History of thyroid disease poorly controlled on prescribed medications
* Use of oral steroids within 30 days prior to screening
* Concurrent medications that are CYP3A4 inducers
* Inability or unwillingness to provide informed consent or abide by the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-11; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of coadministered silymarin and green tea extract at different doses in patients with chronic hepatitis C. | November 2009 to September 2012

SECONDARY OUTCOMES:
To characterize the antioxidant effects of silymarin and EGCG administered alone or in combination. | November 2009 to September 2012

CONTACTS AND LOCATIONS:
Overall Officials: Roy L Hawke, PhD, PharmD, Principal Investigator — UNC School of Pharmacy; Michael W Fried, MD, Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill- UNC Health Care, Chapel Hill, North Carolina, United States